CLINICAL TRIAL: NCT01517308
Title: 24 VS 48-WEEK TREATMENT WITH PEG-IFN ALPHA-2A IN PATIENTS WITH GENOTYPE 2/3 CHRONIC HEPATITIS C, RELAPSERS TO PEG-IFN + RIBAVIRIN TREATMENT. A RANDOMIZED CONTROLLED TRIAL
Brief Title: 24 VS 48-WEEK TREATMENT WITH PEG-IFN ALPHA-2A IN PATIENTS WITH GENOTYPE 2/3 CHRONIC HEPATITIS C
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Time elapsed to require permissions and a recent paper showed a high efficacy of a 48-week regimen in this setting. It seems non-ethical to start this trial
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Prof. Guglielmo Borgia, Full Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.E. Federico II 47/11
Record Dates: First submitted 2012-01-17; First posted 2012-01-25 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Hepatitis C
Keywords: HCV; Hepatitis; Genotype 2 or 3; Pegylated Interferon; Duration
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm 24 weeks (Active Comparator): PEG-IFN α2a 180 μg/week+ ribavirin 800 mg/die for 24 weeks
  Interventions: Drug: pegylated interferon alpha 2a + ribavirin
- Active arm (48 weeks) (Experimental): PEG-IFN α2a 180 μg/week + ribavirin 800 mg/die per 48 weeks
  Interventions: Drug: pegylated interferon alpha 2a + ribavirin

INTERVENTIONS:
Drug: pegylated interferon alpha 2a + ribavirin — Comparison of different duration of drugs (48 weeks vs. 24 weeks)

SUMMARY:
Aim of the present study is to evaluate in a cohort of patients with genotype 2/3 chronic hepatitis C, relapsers to a previous PEG-IFN + ribavirin therapy (alpha-2a or alpha-2b) the efficacy of PEG-IFNα-2a + ribavirin administered for 24 or 48 weeks. It will be evaluated whether 48 weeks of therapy may achieve better results compared to the standard duration (24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age more than 18 years
* Compensated liver disease with following pre-enrollment hematological parameters: Hemoglobin more than 13 g/dl in males and 12 g/dl in females; White blood cell count more than 3,000/mmc; Platelet count more than 100,000 /mmc
* Anti-nuclear antibodies (ANA) less than 1:160
* Anti-Liver-Kidney antibodies (LKM1): negative
* alpha1 fetoprotein levels less than 50 ng/ml in 3 months before enrollment and liver Ultrasound negative for focal malignant lesions.
* HBsAg: negative
* Clinical or histological diagnosis of chronic hepatitis C
* HCV-RNA: positive
* Relapse (end-of-treatment HCV-RNA negativity and positivization within 6 months after therapy withdrawal) to at-least one previous treatment of PEG-IFN (alpha2a or alpha2b) + ribavirin which should have lasted at least for 80% of the 24 planned weeks with at least 80% of total planned dose of PEG-IFN and ribavirin administered.
* Normal values of total and direct bilirubin (with the exception of indirect bilirubin due to extrahepatic factors such as Gilbert syndrome; in these cases the levels should be less than 3 mg/dL).
* Normal values of albumin and creatinin
* Normal fasting glycemia or, in case of glycemic values between 115mg/dL and 140 mg/dl (values confirmed in more than one determination) or if the patient is affected by diabetes mellitus, glycated hemoglobin should be < 8,5%.
* Normal Thyroid Stimulating Hormone (TSH) level. Subjects under pharmacological treatment to maintain normal TSH levels can be enrolled if they fulfill other criteria.
* In case of history of diabetes or hypertension a specialist examination is required to rule out contraindication to therapy.
* Adoption of contraceptive measures

Exclusion Criteria:

* Age less than 18 years
* Women during pregnancy or breast-feeding
* Previous treatment with PEG-IFN alpha2a or alpha2b + ribavirin for more than 6 months
* Participation to any clinical trial within 30 days from enrollment in this protocol
* Subjects with solid organ transplantation (with the exception of cornea or hair transplantation)
* Subject not willing to have a counseling or to abstain from alcohol use
* Suspected hypersensitivity to PEG-Interferon alpha2a or ribavirin
* Any other cause of liver disease different from chronic hepatitis C based on anamnesis of patient or on histological evidence including but not limited to:
* HBV coinfection
* Alpha-1 antitrypsin deficiency
* Wilson disease
* Autoimmune hepatitis
* Alcoholic liver disease
* Hemoglobinopathy included but not limited to thalassemia major.
* Advanced liver diseases diagnosed through history or presence of ascites, esophageal variceal bleeding or hepatic encephalopathy
* Psychiatric conditions: depression or medical history of severe psychiatric alterations such as major psychosis, suicidal ideas, suicidal attempts, depression that required hospitalization or electroconvulsive therapy, prolonged work leave or significant impairment of everyday activities should be excluded. Subjects with history of slight depression might be considered for enrollment in the study if a pre-treatment psychiatric evaluation indicates that the subject is stable and that is possible to follow its mental status during the study.
* Central nervous system trauma or convulsive status requiring treatment.
* Cardiovascular diseases (e.g. angina, congestive heart disease, myocardial infarction, major arrhythmias).
* Decompensated diabetes mellitus
* Clinical gout
* Chronic pulmonary diseases
* Immune-mediated diseases (e.g. chronic inflammatory bowel diseases, idiopathic thrombocytopenic purpura, Systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis)
* Abuse of substances such as alcohol (more than 80 g/die), i.v. or inhalator drugs. Subjects with a history of drug abuse can be enrolled if they were abstinent for at least 2 years.
* Subjects with clinically relevant retinal lesions
* Any other condition that at investigators opinion could be a reason of non suitability for patients or can interfere with his/her participation to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Sustained virological response (SVR) | 6 months after therapy withdrawal
  HCV-RNA undetectability (by the means of Real time PCR assay with a sensitivity limit of 20 UI/mL) 6 months after therapy withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Guglielmo Borgia, Professor, Principal Investigator — Federico II University
Locations (1):
- University of Naples Federico II, Naples, Naples, Italy

REFERENCES:
- [Background] Shiffman ML, Suter F, Bacon BR, Nelson D, Harley H, Sola R, Shafran SD, Barange K, Lin A, Soman A, Zeuzem S; ACCELERATE Investigators. Peginterferon alfa-2a and ribavirin for 16 or 24 weeks in HCV genotype 2 or 3. N Engl J Med. 2007 Jul 12;357(2):124-34. doi: 10.1056/NEJMoa066403. PMID 17625124